CLINICAL TRIAL: NCT05418036
Title: Safety Assessment for Sotalol Protocol in Outpatient Unit
Acronym: Sotalol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Mauricio Ibrahim Scanavacca, Arrhythmia Clinical Unit Director, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4947/19/166
Record Dates: First submitted 2022-06-02; First posted 2022-06-14 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Supraventricular Arrhythmia; Ventricular Arrythmia; Proarrhythmia; Antiarrhythmic Drug Adverse Reaction
Keywords: Sotalol; Drug Safety; Corrected QT interval; Outpatient Treatment
MeSH Terms: interventions — Sotalol

STUDY DESIGN:
Intervention Model Description: Prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Consecutive patients elegible for outpatient sotalol indication (Other): Single Group
  Interventions: Drug: Sotalol Oral Tablet

INTERVENTIONS:
Drug: Sotalol Oral Tablet — Dose of sotalol is prescribed by the attending physician. Accepted for this protocol when the dose is no greater than 160 mg/day
  Other Names: sotalol choridrate

SUMMARY:
Sotalol is an antiarrhythmic medication with proven effects for the suppression and prevention of supraventricular and ventricular arrhythmias. Due to its potential proarrhythmic effect, its introduction should be cautious, and several guidelines recommend starting the medication in hospital settings. However, patients at low risk for a proarrhythmic effect start the medication in outpatient units, despite the lack of clinical studies in the literature that demonstrate the safety of introducing the medication outside the hospital environment.

This research project aims to assess the safety introduction of sotalol in an outpatient unit basis. Our hypothesis is that outpatient introduction of sotalol is safe for low-risk patients and an electrocardiographic analysis after 2 hours of the first dose of medication is a predictor of electrocardiographic changes found after 72 hours.

In this research, serial electrocardiographic analysis with measurements of the QT corrected intervals and its dispersion, as well as clinical and laboratory parameters will be performed in 110 patients.

DETAILED DESCRIPTION:
Participants will be prospectively recruited with sequential electrocardiographic assessments .Their indication and dose will be prescribed at the discretion of the attending physician. The following data to be analyzed are: age, ethnicity, anthropometric data (height, weight and BMI), clinical indication for sotalol, prescribed dose, comorbidities, other concomitant drugs, biochemical analysis (urea, creatinine, estimated creatinine clearance as also sodium, potassium and magnesium serum levels), echocardiogram and Holter monitoring when indicated.

Participants must have a standard 12-lead electrocardiogram (25mm/s) available at the start of treatment, 2 hours after the first dose of medication, and after 3 days, to calculate the corrected QT interval (QTc) and to analyze the dispersion of this interval. The patient will remain in the hospital until the second electrocardiogram is performed.

The QT interval will be measured manually, from the beginning of the QRS to the end of the T wave, by the tangent method, in DII, V5 or V2, in this order of preference. The QTc interval dispersion will be calculated manually, considering the difference between the longest and the shortest QT interval measured in the conventional 12 leads ECG.

All measurements will be made by the same arrhythmologist and later confirmed by a second arrhythmologist. Any divergent measures will be resolved by consensus. If there is no agreement, a third arrhythmologist will analyse the data.

The clinical evolution of the patients (minimum period of 30 days) after the beginning of the medication will be evaluated via face-to-face consultation or by telephone contact. At that moment, the patient's medications, adherence to sotalol use and the occurrence of adverse events will be checked again.

ELIGIBILITY:
Inclusion Criteria:

* Indication of sotalol for the treatment of any supraventricular or ventricular arrhythmias
* Age ≥ 18 years
* Provide written informed consent

Exclusion Criteria:

* Complete bundle branch block
* Bradycardia with a frequency less than or equal to 55 bpm
* Ventricular pacing determined by artificial pacemaker
* Corrected QT interval greater than or equal to 460ms
* Heart failure with reduced ejection fraction, less than 40%
* Lactation period
* Dose required greater than 160 mg/day
* Estimated creatinine clearance less than 60mL/min
* Hypokalemia and hypomagnesemia documented in a patient at risk of spoliation of these components.
* Concomitant use of other drugs with proarrhythmic potential related to increased corrected QT interval (eg, tricyclic antidepressants, macrolide antibiotics, electrolyte-depleting diuretics, etc.).
* Others formal contraindications to the use of sotalol (e.g.: asthma)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Concerns about corrected QT prolongation after 72 hours. | 72 hours from the start of sotalol.
  Number of participants with corrected QT interval increase greater than 10% of the baseline or beyond 500 milliseconds after 72 hours of introduction of sotalol.

SECONDARY OUTCOMES:
Concerns about corrected QT prolongation after 2 hours. | 2 hours after the initiation of sotalol.
  Number of participants with corrected QT interval increase greater than 10% of the baseline or beyond 500 milliseconds after 2 hours of introduction of sotalol.
Side effects that can impair the maintenance of the drug. | 30 days of follow up.
  Side effects that can influence the maintenance of the drug during the 30 days of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio I Scanavacca, MD, PhD, Principal Investigator — Instituto do Coração - HC/FMUSP
Locations (1):
- Clinical Research Center of the Heart Institute - University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh BN. Antiarrhythmic actions of DL-sotalol in ventricular and supraventricular arrhythmias. J Cardiovasc Pharmacol. 1992;20 Suppl 2:S75-90. PMID 1279313
- [Background] Mason JW. A comparison of seven antiarrhythmic drugs in patients with ventricular tachyarrhythmias. Electrophysiologic Study versus Electrocardiographic Monitoring Investigators. N Engl J Med. 1993 Aug 12;329(7):452-8. doi: 10.1056/NEJM199308123290702. PMID 8332150
- [Background] Jurkiewicz NK, Sanguinetti MC. Rate-dependent prolongation of cardiac action potentials by a methanesulfonanilide class III antiarrhythmic agent. Specific block of rapidly activating delayed rectifier K+ current by dofetilide. Circ Res. 1993 Jan;72(1):75-83. doi: 10.1161/01.res.72.1.75. PMID 8417848
- [Background] Sanguinetti MC. Modulation of potassium channels by antiarrhythmic and antihypertensive drugs. Hypertension. 1992 Mar;19(3):228-36. doi: 10.1161/01.hyp.19.3.228. PMID 1548049
- [Background] Sanguinetti MC, Jurkiewicz NK. Two components of cardiac delayed rectifier K+ current. Differential sensitivity to block by class III antiarrhythmic agents. J Gen Physiol. 1990 Jul;96(1):195-215. doi: 10.1085/jgp.96.1.195. PMID 2170562
- [Background] Kehoe RF, Zheutlin TA, Dunnington CS, Mattioni TA, Yu G, Spangenberg RB. Safety and efficacy of sotalol in patients with drug-refractory sustained ventricular tachyarrhythmias. Am J Cardiol. 1990 Jan 2;65(2):58A-64A; discussion 65A-66A. doi: 10.1016/0002-9149(90)90204-e. PMID 2294689
- [Background] Multicentre randomized trial of sotalol vs amiodarone for chronic malignant ventricular tachyarrhythmias. Amiodarone vs Sotalol Study Group. Eur Heart J. 1989 Aug;10(8):685-94. PMID 2676535
- [Background] Obel IW, Jardine R, Haitus B, Millar RN. Efficacy of oral sotalol in reentrant ventricular tachycardia. Cardiovasc Drugs Ther. 1990 Jun;4 Suppl 3:613-8. doi: 10.1007/BF00357039. PMID 2275891
- [Background] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995
- [Background] Neumar RW, Otto CW, Link MS, Kronick SL, Shuster M, Callaway CW, Kudenchuk PJ, Ornato JP, McNally B, Silvers SM, Passman RS, White RD, Hess EP, Tang W, Davis D, Sinz E, Morrison LJ. Part 8: adult advanced cardiovascular life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S729-67. doi: 10.1161/CIRCULATIONAHA.110.970988. PMID 20956224
- [Background] Benditt DG, Williams JH, Jin J, Deering TF, Zucker R, Browne K, Chang-Sing P, Singh BN. Maintenance of sinus rhythm with oral d,l-sotalol therapy in patients with symptomatic atrial fibrillation and/or atrial flutter. d,l-Sotalol Atrial Fibrillation/Flutter Study Group. Am J Cardiol. 1999 Aug 1;84(3):270-7. doi: 10.1016/s0002-9149(99)00275-1. PMID 10496434
- [Background] Prystowsky EN, Benson DW Jr, Fuster V, Hart RG, Kay GN, Myerburg RJ, Naccarelli GV, Wyse DG. Management of patients with atrial fibrillation. A Statement for Healthcare Professionals. From the Subcommittee on Electrocardiography and Electrophysiology, American Heart Association. Circulation. 1996 Mar 15;93(6):1262-77. doi: 10.1161/01.cir.93.6.1262. No abstract available. PMID 8653857
- [Background] January CT, Wann LS, Alpert JS, Calkins H, Cigarroa JE, Cleveland JC Jr, Conti JB, Ellinor PT, Ezekowitz MD, Field ME, Murray KT, Sacco RL, Stevenson WG, Tchou PJ, Tracy CM, Yancy CW; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2014 AHA/ACC/HRS guideline for the management of patients with atrial fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the Heart Rhythm Society. J Am Coll Cardiol. 2014 Dec 2;64(21):e1-76. doi: 10.1016/j.jacc.2014.03.022. Epub 2014 Mar 28. No abstract available. PMID 24685669
- [Background] Knudson JD, Cannon BC, Kim JJ, Moffett BS. High-dose sotalol is safe and effective in neonates and infants with refractory supraventricular tachyarrhythmias. Pediatr Cardiol. 2011 Oct;32(7):896-903. doi: 10.1007/s00246-011-0010-0. Epub 2011 May 8. PMID 21553267
- [Background] van der Heijden LB, Oudijk MA, Manten GT, ter Heide H, Pistorius L, Freund MW. Sotalol as first-line treatment for fetal tachycardia and neonatal follow-up. Ultrasound Obstet Gynecol. 2013 Sep;42(3):285-93. doi: 10.1002/uog.12390. PMID 23303470
- [Background] Jaeggi ET, Carvalho JS, De Groot E, Api O, Clur SA, Rammeloo L, McCrindle BW, Ryan G, Manlhiot C, Blom NA. Comparison of transplacental treatment of fetal supraventricular tachyarrhythmias with digoxin, flecainide, and sotalol: results of a nonrandomized multicenter study. Circulation. 2011 Oct 18;124(16):1747-54. doi: 10.1161/CIRCULATIONAHA.111.026120. Epub 2011 Sep 19. PMID 21931080
- [Background] Hill GD, Kovach JR, Saudek DE, Singh AK, Wehrheim K, Frommelt MA. Transplacental treatment of fetal tachycardia: A systematic review and meta-analysis. Prenat Diagn. 2017 Nov;37(11):1076-1083. doi: 10.1002/pd.5144. PMID 28833310
- [Background] Lopes NH, Grupi C, Dina CH, de Gois AF, Hajjar LA, Ayub B, Rochitte CE, Ramires JA, Hueb WA, Kalil R. [QT interval dispersion analysis in acute myocardial infarction patients: coronary reperfusion effect]. Arq Bras Cardiol. 2006 Aug;87(2):91-8. doi: 10.1590/s0066-782x2006001500005. Portuguese. PMID 16951825
- [Background] Wolbrette DL. Risk of proarrhythmia with class III antiarrhythmic agents: sex-based differences and other issues. Am J Cardiol. 2003 Mar 20;91(6A):39D-44D. doi: 10.1016/s0002-9149(02)03378-7. PMID 12670641
- [Background] Shantsila E, Watson T, Lip GY. Drug-induced QT-interval prolongation and proarrhythmic risk in the treatment of atrial arrhythmias. Europace. 2007 Sep;9 Suppl 4:iv37-44. doi: 10.1093/europace/eum169. PMID 17766322
- [Background] Weeke P, Delaney J, Mosley JD, Wells Q, Van Driest S, Norris K, Kucera G, Stubblefield T, Roden DM. QT variability during initial exposure to sotalol: experience based on a large electronic medical record. Europace. 2013 Dec;15(12):1791-7. doi: 10.1093/europace/eut153. Epub 2013 Jun 19. PMID 23787903
- [Background] Pratt CM, Camm AJ, Cooper W, Friedman PL, MacNeil DJ, Moulton KM, Pitt B, Schwartz PJ, Veltri EP, Waldo AL. Mortality in the Survival With ORal D-sotalol (SWORD) trial: why did patients die? Am J Cardiol. 1998 Apr 1;81(7):869-76. doi: 10.1016/s0002-9149(98)00006-x. PMID 9555777
- [Background] Sullivan SD, Orme ME, Morais E, Mitchell SA. Interventions for the treatment of atrial fibrillation: a systematic literature review and meta-analysis. Int J Cardiol. 2013 May 10;165(2):229-36. doi: 10.1016/j.ijcard.2012.03.070. Epub 2012 Apr 1. PMID 22469557
- [Background] Lafuente-Lafuente C, Valembois L, Bergmann JF, Belmin J. Antiarrhythmics for maintaining sinus rhythm after cardioversion of atrial fibrillation. Cochrane Database Syst Rev. 2015 Mar 28;(3):CD005049. doi: 10.1002/14651858.CD005049.pub4. PMID 25820938
- [Background] Coughtrie AL, Behr ER, Layton D, Marshall V, Camm AJ, Shakir SAW. Drugs and life-threatening ventricular arrhythmia risk: results from the DARE study cohort. BMJ Open. 2017 Oct 16;7(10):e016627. doi: 10.1136/bmjopen-2017-016627. PMID 29042382
- [Background] Finks SW, Rogers KC, Manguso AH. Assessment of sotalol prescribing in a community hospital: opportunities for clinical pharmacist involvement. Int J Pharm Pract. 2011 Aug;19(4):281-6. doi: 10.1111/j.2042-7174.2011.00094.x. Epub 2011 Mar 15. PMID 21733016
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Halperin JL, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Tamargo JL, Zamorano JL; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines; European Heart Rhythm Association; Heart Rhythm Society. ACC/AHA/ESC 2006 Guidelines for the Management of Patients with Atrial Fibrillation: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation): developed in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. Circulation. 2006 Aug 15;114(7):e257-354. doi: 10.1161/CIRCULATIONAHA.106.177292. No abstract available. PMID 16908781
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Priori SG, Blomstrom-Lundqvist C, Mazzanti A, Blom N, Borggrefe M, Camm J, Elliott PM, Fitzsimons D, Hatala R, Hindricks G, Kirchhof P, Kjeldsen K, Kuck KH, Hernandez-Madrid A, Nikolaou N, Norekval TM, Spaulding C, Van Veldhuisen DJ; ESC Scientific Document Group. 2015 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: The Task Force for the Management of Patients with Ventricular Arrhythmias and the Prevention of Sudden Cardiac Death of the European Society of Cardiology (ESC). Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC). Eur Heart J. 2015 Nov 1;36(41):2793-2867. doi: 10.1093/eurheartj/ehv316. Epub 2015 Aug 29. No abstract available. PMID 26320108
- [Background] Agusala K, Oesterle A, Kulkarni C, Caprio T, Subacius H, Passman R. Risk prediction for adverse events during initiation of sotalol and dofetilide for the treatment of atrial fibrillation. Pacing Clin Electrophysiol. 2015 Apr;38(4):490-8. doi: 10.1111/pace.12586. Epub 2015 Jan 28. PMID 25626340
- [Background] Sauer AJ, Kaplan R, Xue J, Dorsey P, Hayes M, Shah SJ, Passman R. Electrocardiographic markers of repolarization heterogeneity during dofetilide or sotalol initiation for paroxysmal atrial fibrillation. Am J Cardiol. 2014 Jun 15;113(12):2030-5. doi: 10.1016/j.amjcard.2014.03.047. Epub 2014 Apr 1. PMID 24793679